CLINICAL TRIAL: NCT06875908
Title: Reliability and Validity of the Turkish Version of General Sleep Disturbance Scale (GSDS-T) in Multiple Sclerosis
Status: Recruiting | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Emel Mete, Assistant Professor, PhD, Istanbul Medeniyet University
Other Study IDs: MS-GSDS
Record Dates: First submitted 2025-03-09; First posted 2025-03-13 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis; Sleep Disturbance
Keywords: Multiple sclerosis; Sleep disturbances
MeSH Terms: conditions — Multiple Sclerosis; Parasomnias

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with MS: Turkish Validity and Reliability of The GSDS-T in patients with multiple sclerosis The aim of this study is to investigate the validity and reliability of the Turkish version of general sleep disturbance scale (GSDS-T) in patients with multiple sclerosis. It has 21 questions. This study will be conducted on patients with multiple sclerosis. In order to evaluate the validity of the GSDS-T, the Pittsburgh Sleep Quality Index (PSQI) which can evaluate sleep quality and has been validated in Turkish, will be used. Scales will be repeated after 15 days to assess test-retest reliability.
  Interventions: Other: Turkish Validity and Reliability of The GSDS-T in patients with multiple sclerosis

INTERVENTIONS:
Other: Turkish Validity and Reliability of The GSDS-T in patients with multiple sclerosis — The aim of this study is to investigate the validity and reliability of the Turkish version of general sleep disturbance scale (GSDS-T) in patients with multiple sclerosis. It has 21 questions. This study will be conducted on patients with multiple sclerosis. In order to evaluate the validity of the GSDS-T, the Pittsburgh Sleep Quality Index (PSQI) which can evaluate sleep quality and has been validated in Turkish, will be used. Scales will be repeated after 15 days to assess test-retest reliability.

SUMMARY:
The GSDS-T was developed by Lee KA to assess difficulty falling asleep, waking up during sleep, sleep quality, and daytime alertnes. The Turkish validity and reliability of the scale have been conducted on stroke patients but not on multiple sclerosis patients. The aim of this study is to investigate the validity and reliability of the Turkish version of general sleep disturbance scale (GSDS-T) in patients with multiple sclerosis

DETAILED DESCRIPTION:
The GSDS-T was developed by Lee KA to assess difficulty falling asleep, waking up during sleep, sleep quality, and daytime alertnes. The Turkish validity and reliability of the scale has been conducted on stroke patients but not on multiple sclerosis patients. The aim of this study is to investigate the validity and reliability of the Turkish version of general sleep disturbance scale (GSDS-T) in patients with multiple sclerosis. GSD has 21 questions. This study will be conducted on patients with multiple sclerosis (MS). 126 participants will be included in the study. In order to evaluate the validity of the GSDS-T, the Pittsburgh Sleep Quality Index (PSQI) which can evaluate sleep quality and has been validated in Turkish, will be used. Scales will be repeated after 15 days to assess test-retest reliability.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over the age of 18 who have been diagnosed with Multiple Sclerosis for at least two years,
* Those with an EDSS score >2.
* Those without symptoms of insomnia according to the Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) diagnostic criteria
* Individuals whose native language is Turkish and who have the ability to speak and understand.

Exclusion Criteria:

* Those with severe spasticity,
* Those with vision and hearing problems,
* Those with a known mental illness (major depression, schizophrenia, psychosis, etc.),
* Those in an acute relapse phase,
* Those using dietary supplements,
* Those using tranquilizers or immunosuppressants.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Multiple sclerosis who are aged 18-65 years with EDSS score > 2 and able to speak and read Turkish.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-07-20 (Estimated); Study Completion 2025-08-10 (Estimated)

PRIMARY OUTCOMES:
Sleep disturbances | baseline
  Sleep disturbances will be assessed with the general sleep disturbance scale (GSDS). It consists of 21 items in total. Each item is scored on a scale of 0-7 includes six sub-categories: Difficulty falling asleep, waking up from sleep; sleep quality; sleep duration; daytime sleepiness; and taking supplements to help sleep. The total score is the calculated sum of 21 items. The minimum score is "0" while the maximum score is "147" points. Higher scores indicate more sleep disturbances.
Sleep quality | baseline
  Sleep quality will be assessed with the Pittsburgh Sleep Quality Index (PSQI). The PSQI consists of 24 questions in total. The scale has 7 components: sleep quality (component 1), sleep latency (component 2), sleep duration (component 3), habitual sleep efficiency (component 4), sleep disturbance (component 5), use of sleeping pills (component 6), and daytime sleep dysfunction (component 7). Each component is evaluated on a 0-3 scale. The sum of these 7 component scores gives the total PSQI score. The total PSQI score varies between 0-21. While the sleep quality of individuals with a total score of 5 and below is evaluated as "good," the sleep quality of individuals with a score above 5 is evaluated as "poor."

CONTACTS AND LOCATIONS:
Locations (1):
- Bağcılar Training and Research Hospital, Bağcılar, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No